CLINICAL TRIAL: NCT06589401
Title: A Phase I Trial Evaluating the Safety, Tolerability, and Pharmacokinetic Profile of INP12 in Patients with Advanced Solid Tumors
Brief Title: Oral Paclitaxel for Patients with Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: InnoUp Farma S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INP12-01
Record Dates: First submitted 2023-06-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor
Keywords: Oral paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- INP12 (Experimental): In Part A (dose escalation), INP12 will be administered for 3 consecutive weeks (Days 1, 8, and 15) based on 28-day cycles. At least 3 patients will be included in each dose level. Each patient will be evaluated for dose-limiting toxicity (DLT) throughout the first cycle (28 days).
  In Part B (dose expansion), once the MTD is reached (or the highest protocol-defined dose in the absence of exceeding the MTD), an expanded cohort will be evaluated with the dose level of the MTD, or an intermediate one.
  Interventions: Drug: INP12

INTERVENTIONS:
Drug: INP12 — Oral paclitaxel

SUMMARY:
Phase I trial evaluating the safety, tolerability, and pharmacokinetic profile of INP12, a nanoparticles-based oral paclitaxel, in patients with advanced solid tumors

The aim in Part A (Escalation phase) is to determine the maximum tolerated dose (MTD) or the highest protocol-defined dose (in the absence of exceeding the MTD)and the recommended phase II dose (RP2D) of INP12 administered orally once a week during three consecutive weeks under a 28-day cycle in patients with advanced solid tumors.

The aim in Part B (Expansion phase) is to assess the safety and tolerability of INP12 as monotherapy at the RP2D or highest protocol-defined dose in patients with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients; age ≥ 18 years at the time of study entry.
* Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.

Part A: Patients with a histologically and/or cytological confirmed solid tumor that is advanced and/or metastatic.

Part B: Patients with a histologically and/or cytological confirmed solid tumor that is advanced and/or metastatic from which at least 50% should be patients with advanced or metastatic breast cancer.

*Note: If at the beginning of the phase-expansion there are patients still receiving INP12 in the phase-escalation, they will be offered to continue treatment with INP12 at the dose defined for the expansion phase.

* Patients for which standard therapy does not exist or is no longer effective.
* ECOG ≤ 2.
* Life expectancy of at least 12 weeks.
* No previous treatment with growth factors or blood transfusions within 28 days prior to the first dose of INP12.
* Patient with adequate organ and spinal function:

  * Absolute neutrophil count (ANC) ≥ 1500/mm3
  * Hemoglobin ≥ 9 g/dL
  * Platelets (PTL) ≥ 100,000 mm3
  * Alanine aminotransferase (ALT) / aspartate aminotransferase (AST) ≤ 2.5 x upper limit normal (ULN) (≤ 5 x ULN in case of hepatocellular carcinoma [HHC] or liver metastases)
  * Total bilirubin ≤ 1.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or Creatinine clearance ≥ 50 mL/min (Cockcroft and Gault formula)
* Patient with measurable or evaluable lesion.
* Females of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception from the time of screening and must agree to continue using such precautions for 90 days after the last dose of investigational product. Male partners of a female patient must use male condom plus spermicide throughout this period. * A woman is considered to be of childbearing potential from menarche to postmenopausal unless permanently sterilized. Sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menstruation for 12 months without an alternative medical cause. According to the CTFG recommendations, are considered highly effective contraceptive methods**: Combined hormonal treatment containing estrogen and progestogen (oral, intravaginal, transdermal); progestogen hormonal contraception associated with ovulation inhibition (oral, injectable, implantable); intrauterine device (IUD), hormone-releasing intrauterine system (IUS); bilateral tubal occlusion; vasectomized partner; sexual abstinence.
* Unsterilized and sexually active men who have a fertile female partner should use 2 effective and acceptable contraceptive methods from day 1 up to 90 days after receiving the last dose of INP12. Periodic abstinence, rhythm method, and interrupted intercourse are not acceptable contraceptive methods.
* Patients available for periodic blood tests and evaluations related to the study.
* Patients able and willing to comply with study procedures as per protocol.

Exclusion Criteria:

* Simultaneous enrollment in another clinical study unless it is an observational (non-interventional) study or the follow-up period of an interventional study.
* History of severe allergic reactions (ie, Grade 4 allergy, anaphylactic reaction from which the patient did not recover within 6 hours of institutional supportive care) to an unknown allergen or any components of the study drug formulations.
* Patients with dysphagia or disorders in gastrointestinal function.
* Previous hypersensitive reaction to taxanes.
* Previous hypersensitive reaction to corn.
* Concomitant systemic chemotherapy, hormonal therapy, and immunotherapy for the treatment of cancer.
* The concomitant use of hormones for non-oncological diseases is acceptable (eg, insulin for diabetes and hormone replacement therapy). Concurrent use of hormones for non-cancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable.
* Local treatment of isolated lesions with palliative intent is acceptable (eg, through surgery or local radiotherapy).
* Concomitant use of cytochrome P-450 (CYP) 3A4 inhibitors and/or inducers.
* Concomitant use of P-glycoprotein 1 (Pgp) inhibitors and/or inducers.
* Previous or current use of immunosuppressive drugs ≤ 28 days prior to the first dose of INP12, except intranasal, topical, and inhaled corticosteroids.
* Receipt of any conventional or investigational anticancer therapy not otherwise specified above within 28 days prior to the first dose of INP12.
* Primary central nervous system (CNS) tumor or untreated CNS metastatic disease, including leptomeningeal disease or spinal cord compression, except for previously treated patients who are asymptomatic and who have not required corticosteroids (at any dose) or anticonvulsants for at least 14 days before the selection.
* History of malignant tumors in the last 2 years, except for malignant non-invasive neoplasms, such as cervical carcinoma in situ, non-melanoma skin carcinoma, or ductal carcinoma in situ of the breast, cured by surgery.
* Unresolved AEs from a previous cancer treatment, defined according to the NCI CTCAE v5.0 classification (see Appendix 15.1) as unresolved events up to grade 0 or 1, or up to the levels required in the inclusion/exclusion criteria, with the exception of alopecia and laboratory values listed per the inclusion criteria Patients with irreversible toxicity that is not reasonably expected to be exacerbated by any of the investigational products may be included (eg, hearing loss).
* Pregnant or breastfeeding women.
* Patients with a known HIV infection, chronic or active hepatitis B or C or active hepatitis A.
* Patients with difficulty in swallowing or with any disorder in the gastrointestinal system that may affect the intake and/or absorption of the study drug.
* Major surgery (as defined by the Investigator) within 4 weeks prior to first dose of INP12 or still recovering from prior surgery. Local surgery of isolated lesions for palliative intent is acceptable.
* Severe or uncontrolled medical condition including but not limited to ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer, intense gastritis, or psychiatric disorder/social situations that limit compliance with the protocol.
* Any condition that, according to the Investigator, could potentially hamper compliance with the study protocol, the evaluation of INP12, the interpretation of the patient's safety, the study results, or the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
• MTD determination | 28 days
  To determine the maximum tolerated dose (MTD) or the highest protocol-defined dose (in the absence of exceeding the MTD) and the recommended phase II dose (RP2D) of INP12 administered orally once weekly in patients with advanced solid tumors.
• Incidence of INP12 Adverse Events (Safety and tolerability profile of INP12) | 28 days
  Tolerability will be defined by the number of patients experiencing any dose limiting toxicity (DLT) during the first 28-day cycle of INP12.
  Safety of INP12 will be assessed on the incidence rate, severity, and relationship to treatment of adverse events (AEs) and serious adverse events (SAEs) according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) V4.03 (see Appendix 15.2).
  Other assessments will include safety laboratory parameters, vital signs, and electrocardiograms (ECG) in each dose group and in the expansion phase.

CONTACTS AND LOCATIONS:
Locations (1):
- VHIO, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No